CLINICAL TRIAL: NCT01370473
Title: Institutional Registry of Hyponatremia
Acronym: Hyponatremia
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1050
Record Dates: First submitted 2011-05-02; First posted 2011-06-10 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Hyponatremia
Keywords: Hyponatremia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to create an institutional and population-based registry of Hyponatremia with a prospective survey based on epidemiological data, risk factors, diagnosis, prognosis, treatment, monitoring and survival.

This study will also describe the occurrence of hyponatremia in the population of HIBA in the Central Hospital, as well as the characteristics of clinical presentation, evolution and predisposing factors of hyponatremia.

DETAILED DESCRIPTION:
Alterations in plasma sodium concentration (sodium ratio and solvent) are very common in clinical practice. Since plasma sodium concentration is a major determinant of plasma osmolality, it will determine the balance of the different body fluids compartments.

Hyponatremia is defined as the measurement of plasma sodium below 136 mmol per liter. Hyponatremia may be associated with normal tone, low or high. The pseudohyponatremia is an artifact of measuring the concentration of sodium in the context of a growth in the concentration of active osmoles (glucose, mannitol), which induce water movement from the intracellular to extracellular. This can also occur in the context of substances that do not generate osmolarity as triglycerides and plasma proteins. In the first case, the investigators are in the presence of hypertonic hyponatremia, in the second case to an isotonic hyponatremia, neither should be considered true hyponatremias.

The hypotonic hyponatremia is the one considered to be true. It represents the most common electrolyte imbalance in hospitalized patients (2% to 22% depending on the series and the cutoff points) and outpatients (7% to 18% in tertiary care center, being very dependent variable and cutoffs series). It is associated with increased morbidity and mortality (18% in hospitalized patients). It can be the cause of serious illness that requires immediate attention or be a marker of morbidity and mortality for underlying diseases (congestive heart failure, liver cirrhosis).

Hyponatremia can occur in a wide range of patients, from asymptomatic with good tolerance to the critically ill. Symptoms may be mild or severe, and none is specific. They are mainly neurological and generally reflect dysfunction associated with cerebral edema. They are caused due to the magnitude of the alteration of plasma sodium concentration and the system speed.

The clinical management challenge is the identification and specific treatment of the cause, understanding that the study of it brings the knowledge of its pathophysiology. The latter can be grouped into a loss of sodium and / or gain of fluid. In turn, the gain of liquids is possible by an alteration in kidney dilusorios mechanisms, as well as the variations that according to the glomerular filtration rate and filtered sodium load. Its high prevalence and potential neurologic sequelae associated with the disease and its treatment make the diagnosis and appropriate treatment is mandatory. Traditionally, the initial assessment and treatment are suboptimal in the descriptive series.

We have not found in the literature any systematic record of patients with abnormalities in the sodium concentration in both inpatients and outpatients, except for a record of pharmacological effects. We believe that while this is a highly prevalent disorder, is not attractive to the pharmaceutical industry and this would partly explain the apparent lack of studies with large groups of patients.

We also have not found any descriptive studies conducted in Argentina. While there are multiple proposals for the evaluation of alterations in sodium, there is no standardization in our single on the cleavage of specific sodium, appropriate diagnostic evaluation and proposed the best treatment for hyponatremia. There are technical difficulties in the standardization of the assessment of symptoms, physical examination, and the effectiveness of clinical parameters to guide therapy.

There are no reports of the strategy used in our country for diagnosis and decision making in patients with alterations of plasma sodium concentrations. Nor Disnatremias epidemiological data in our environment, risk factors, assessment and monitoring of survival, complications and recurrences. We have no references in the literature that talk about the behaviour of the disnatremias in the areas of inpatient and outpatient, there are no data to see whether treatments aimed at the mere correction of hyponatremia, or interpretation of the pathophysiological same.

The systematic recording of cases of Disnatremias will reveal the characteristics of the disease in our environment, the diagnostic strategies used and their results and the time course of the disease. We believe that this knowledge will allow us to design studies to optimize and standardize the diagnostic strategies, evaluation and treatment, resulting in a benefit for the affected population.

ELIGIBILITY:
Inclusion Criteria:

1. Over 17 years.
2. At least a measure of central laboratory Na less than 130 mmol / l in patients without criteria for chronic hyponatremia or at least a measure of central laboratory Na greater than or equal to 150 mmol / l.
3. First detection of sodium less than 130 mmol / l defined as exacerbation of chronic hyponatremia patients.
4. Reepisodio defined as hyponatremia in patients who recovered the acute episode and again have a new episode of acute hyponatremia.

Exclusion Criteria:

1. The refusal to register or to the informed consent process.
2. Error in the measurement of sodium in the opinion of treating physician / recognized laboratory.
3. Chronic renal patients on hemodialysis or peritoneal dialysis.
4. Sodium determinations patients with cardiovascular surgery during cardiopulmonary bypass with intraoperative sodium determinations.
5. Outpatients (excluding patients with PS on guard and spontaneous demand, see definitions).
6. Patients treated (removal of blood and determination of serum sodium) in San Justo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with hyponatremia
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2006-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
clinical features | feature clinics are evaluated during the acute episode and mortality were measured in the acute episode and in the semiannual monitoring by telephone
  Signs and symptoms Hospital Length of Stay Mortality Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Giunta, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina